CLINICAL TRIAL: NCT01135719
Title: A Prospective Randomized Comparison of Fellow Eyes Undergoing LASIK or PRK With a Wavefront-guided Excimer Laser Versus a Wavefront-optimized Excimer Laser
Brief Title: A Comparison of Fellow Eyes Undergoing LASIK or PRK With a Wavefront-guided Excimer Laser Versus a Wavefront-optimized Excimer Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward E. Manche (Other)
Responsible Party: Sponsor-Investigator, Edward E. Manche, Stanford University School of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-04302009-2458
Record Dates: First submitted 2009-05-08; First posted 2010-06-03 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Hyperopia; Myopia; Astigmatism
Keywords: Myopia; Hyperopia; Astigmatism; PRK; LASIK
MeSH Terms: conditions — Hyperopia; Myopia; Astigmatism | interventions — Keratomileusis, Laser In Situ; Photorefractive Keratectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wavefront guided LASIK/PRK (Active Comparator): Wavefront-guided LASIK/PRK
  Interventions: Procedure: LASIK and PRK
- Wavefront optimized LASIK/PRK (Active Comparator): Wavefornt optimized LASIK/PRK
  Interventions: Procedure: LASIK and PRK

INTERVENTIONS:
Procedure: LASIK and PRK — Wavefront-guided versus wavefront-optimized LASIK or PRK.
  Other Names: Allegretto Wave Eye-Q 400 Hz excimer laser; Visx CustomVue excimer laser; Laser in-situ keratomileusis; Photorefractive keratectomy; Wavefront-guided; Wavefront-optimized

SUMMARY:
Subjects with myopia, hyperopia and astigmatism are being randomized to be treated in one eye with a wavefront-guided excimer laser and their fellow eye treated with a wavefront-optimized excimer laser.

DETAILED DESCRIPTION:
Subjects with myopia, hyperopia and astigmatism are being randomized by ocular dominance to be treated with either PRK or LASIK. One eye will be treated with a wavefront-guided excimer laser and the fellow eye will be treated with a wavefront optimized excimer laser.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects age 21 and older.
* Subjects with nearsightedness, farsightedness and/or astigmatism.

Exclusion Criteria:Autoimmune diseases.

* Children.
* Women pregnant or nursing.
* Ectatic corneal disease.
* Previous ocular surgery.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Changes in best spectacle corrected visual acuity. | One year
Changes in 25 and 5% low contrast visual acuity. | One year
Improvement in uncorrected visual acuity | One year

SECONDARY OUTCOMES:
Changes in higher order aberrations. | One year
Topographic changes. | One year
Quality of vision changes. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Edward E. Manche, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Smith RG, Manche EE. One-Year Outcomes From a Prospective, Randomized, Eye-to-Eye Comparison of Wavefront-Guided and Wavefront-Optimized PRK in Myopia. J Refract Surg. 2020 Mar 1;36(3):160-168. doi: 10.3928/1081597X-20200129-01. PMID 32159820
- [Background] Lee MD, Toy BC, Manche EE. Astigmatic outcomes in myopic wavefront-guided laser in situ keratomileusis versus wavefront-guided photorefractive keratectomy using vector analysis. J Cataract Refract Surg. 2018 Nov;44(11):1350-1354. doi: 10.1016/j.jcrs.2018.07.022. Epub 2018 Sep 7. PMID 30201128
- [Background] He L, Manche EE. Contralateral eye-to-eye comparison of wavefront-guided and wavefront-optimized photorefractive keratectomy: a randomized clinical trial. JAMA Ophthalmol. 2015 Jan;133(1):51-9. doi: 10.1001/jamaophthalmol.2014.3876. PMID 25321951
- [Background] Kung JS, Manche EE. Quality of Vision After Wavefront-Guided or Wavefront-Optimized LASIK: A Prospective Randomized Contralateral Eye Study. J Refract Surg. 2016 Apr;32(4):230-6. doi: 10.3928/1081597X-20151230-01. PMID 27070229
- [Background] He L, Liu A, Manche EE. Wavefront-guided versus wavefront-optimized laser in situ keratomileusis for patients with myopia: a prospective randomized contralateral eye study. Am J Ophthalmol. 2014 Jun;157(6):1170-1178.e1. doi: 10.1016/j.ajo.2014.02.037. Epub 2014 Feb 19. PMID 24560995
- [Background] Sales CS, Manche EE. One-year eye-to-eye comparison of wavefront-guided versus wavefront-optimized laser in situ keratomileusis in hyperopes. Clin Ophthalmol. 2014 Nov 12;8:2229-38. doi: 10.2147/OPTH.S70145. eCollection 2014. PMID 25419115